CLINICAL TRIAL: NCT05339724
Title: Platelets: A Neglected Cell in Cystic Fibrosis Lung Inflammation
Brief Title: Platelets in Cystic Fibrosis Lung Inflammation
Status: Completed | Type: Observational
Sponsor: Mersin Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ali Özdemir, Assoc Prof, Mersin Training and Research Hospital
Other Study IDs: 2022/138
Record Dates: First submitted 2022-04-08; First posted 2022-04-21 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Platelet Levels and Mean Platelet Volume in Patients With CF
Keywords: cystic fibrosis, platelet count, mean platelet volume
MeSH Terms: conditions — Cystic Fibrosis | interventions — Platelet Count

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group 1. Total cystic fibrosis patients with pulmonary exacerbation: Platelet count (PC) and mean platelet volume (MPV) during pulmonary exacerbation.
  Interventions: Other: platelet count and mean platelet volume are obtained from whole blood count
- Group 2. Total cystic fibrosis patients with no pulmonary exacerbation: PC and MPV during no pulmonary exacerbation
  Interventions: Other: platelet count and mean platelet volume are obtained from whole blood count
- Group 3. Cystic fibrosis patients with chronic colonization in acute pulmonary exacerbation: PC and MPV during chronic colonization in acute pulmonary exacerbation
  Interventions: Other: platelet count and mean platelet volume are obtained from whole blood count
- Group 4. Cystic fibrosis patients with chronic colonization without pulmonary exacerbation: PC and MPV during chronic colonization without pulmonary exacerbation
  Interventions: Other: platelet count and mean platelet volume are obtained from whole blood count
- Group 5. Cystic fibrosis patients with chronic colonization without pulmonary exacerbation: PC and MPV during chronic colonization without pulmonary exacerbation
  Interventions: Other: platelet count and mean platelet volume are obtained from whole blood count
- Group 6. Cystic fibrosis patients with no chronic colonization without pulmonary exacerbation: PC and MPV during no chronic colonization without pulmonary exacerbation
  Interventions: Other: platelet count and mean platelet volume are obtained from whole blood count

INTERVENTIONS:
Other: platelet count and mean platelet volume are obtained from whole blood count — The records of cystic fibrosis patients will be retrospectively evaluated for acute pulmonary exacerbation, chronic airway colonization for bacteria, clinical stable status. PC and MPV will be obtained and matched in 6 groups (described above). Then, PC and MPV will be compared among the groups.

SUMMARY:
Cystic fibrosis (CF) is a chronic multiorgan disorder caused by mutations in the CFTR (cystic fibrosis transmembrane conductance regulator) gene. Chronic airway infection by bacterial pathogens accounts for the progressive, suppurative pulmonary disease that leads to significant morbidity and mortality in patients with CF. Neutrophil recruitment to the lungs accounts the most important contributor to pulmonary destruction. However, there is evidence that platelets may also have an important role in the pathogenesis of inflammation. To our knowledge, there is few information in platelet levels in patients with cystic fibrosis during pulmonary exacerbation, chronic airway colonization and when stable.

DETAILED DESCRIPTION:
Airway inflammation in CF is predominantly neutrophilic in nature with increased concentrations of pro-inflammatory mediators include TNF-α, IL-1β, IL-6, IL-8, IL-17, IL-33, GM-CSF and G-CSF. In addition, other cell types including macrophages and T-lymphocytes are expressed by CFTR and contribute to the CF inflammatory response.

Researches have indicated that platelets may also have a significant contribution to the inflammation. Platelet depletion or antiplatelet therapies attenuate injury and mortality in animal models of acute lung injury. More importantly, CFTR expression has been shown on human platelets. Recent data suggests that CF patients have an increase in circulating activated platelets and platelet reactivity.

Taken together, these observations support a potentially important role of platelets in regulating lung inflammation in CF. However, there are few studies examine platelet and lung inflammation interraction in patients with CF. Therefore we aimed to investigate platelet count (PC) and mean platelet volume (MPV) levels in various conditions in our CF patients.

ELIGIBILITY:
Inclusion Criteria:

* All regularly followed cystic fibrosis patients with clinical and laboratory results could be obtained from medical charts.

Exclusion Criteria:

* None

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cystic fibrosis patients
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Platelet levels and mean platelet volume in acute pulmonary infection in patients with cystic fibrosis | 2 weeks
  Elevated platelet level count (x103/uL) and increased mean platelet volume (fl) during acute pulmonary exacerbation in cystic fibrosis patients

CONTACTS AND LOCATIONS:
Overall Officials: Ali Özdemir, MD, Principal Investigator — Assoc Prof, Mersin City Research & Training Hospital; Murat Ersoy, MD, Study Chair — Clinical Pediatrician, Mersin City Research & Training Hospital
Locations (1):
- Mersin City Research & Training Hospital, Mersin, Turkey (Türkiye)